CLINICAL TRIAL: NCT04474145
Title: The Effect of Combined Hydrodilatation, Corticosteroid Injection, and Joint Mobilization for Treament of Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20191212R; NSTC 109-2314-B-341-002 (Other Grant/Funding Number: National Science and Technology Council); NSTC 110-2314-B-341-002 (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Frozen Shoulder; Hydrodilatation; Joint Mobilization; Corticosteroid Injection; Physical Therapy; Rehabilitation
Keywords: frozen shoulder; hydrodilatation; joint mobilization; corticosteroid injection; physical therapy; rehabilitation
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comb group (Active Comparator): Patients in the Comb group will receive hydrodilatation of the affected shoulder and subdeltoid bursa injection for 2 times in 2-week interval. Patients also receive mobilization exercise and conventional physical therapy (including physical modalities and stretch exercise), 3 times a week, for 8 weeks.
  The injectates for hydrodilation include 10mg triamcinolone, 2cc 1% xylocaine, and 17cc normal saline for both posterior and anterior shoulder joint injection. 10mg triamcinolone and 2cc 1% xylocaine will also be injected into the subdeltoid bursa of the affected shoulder. All injections will be performed under ultrasound guidance. For shoulder joint injection, ａ21 gauge, 3-inch needle will be used; and a 22 gauge, 1.5 inch needle will be applied for subdeltoid bursa injection.
  Interventions: Procedure: Comb group
- PT group (Active Comparator): The physiotherapy program includes physical modalities (heat therapy and electric therapy) and therapeutic exercise (stretching, ROM exercise, and strengthening), three times a week, and will be continued for 8 weeks or until total recovery of the symptoms. The stretching exercise program is similar to the stretching exercise described above. For mimicking injection in the Comb group, patients in the PT group will receive 2cc 1% xylocain injection at the posterior deltoid muscle.
  Interventions: Procedure: PT group

INTERVENTIONS:
Procedure: Comb group — Patients in the Comb group will receive hydrodilatation of the affected shoulder and subdeltoid bursa injection for 2 times in 2-week interval. Patients also receive mobilization exercise and conventional physical therapy (including physical modalities and stretch exercise), 3 times a week, for 8 weeks.
  The injectates for hydrodilation include 10mg triamcinolone, 2cc 1% xylocaine, and 17cc normal saline for both posterior and anterior shoulder joint injection. 10mg triamcinolone and 2cc 1% xylocaine will also be injected into the subdeltoid bursa of the affected shoulder. All injections will be performed under ultrasound guidance. For shoulder joint injection, ａ21 gauge, 3-inch needle will be used; and a 22 gauge, 1.5 inch needle will be applied for subdeltoid bursa injection.
  Arms: Comb group
Procedure: PT group — The physiotherapy program includes physical modalities (heat therapy and electric therapy) and therapeutic exercise (stretching, ROM exercise, and strengthening), three times a week, and will be continued for 8 weeks or until total recovery of the symptoms. The stretching exercise program is similar to the stretching exercise described above. For mimicking injection in the Comb group, patients in the PT group will receive 2cc 1% xylocain injection at the posterior deltoid muscle.
  Arms: PT group

SUMMARY:
The effect of combination of hydrodilatation, corticosteroid injection, and joint mobilization for treatment of frozen shoulder, compared with general physical therapy.

DETAILED DESCRIPTION:
Frozen shoulder (FS) is a common clinical problem which induces pain, loss of passive and active range of motion (ROM) of glenohumeral joint, and leads to disability, functional limitation, and decreasing quality of life. FS is usually treated with conservative treatments, which include medications, physiotherapy, joint mobilization, hydrodilatation, intra-articular steroid injection, etc.. The short-term effect of each treatment is variable, and the long-term effect is not established. Clinically combination of each treatment is common, but types of combination, and the effect of combination is still not well studied. We aim to combine hydrodilatation (with corticosteroid injection), joint mobilization, and general physiotherapy to treat frozen shoulder and compare the long-term effect with general physical therapy alone.

This is a prospective single-blind randomized controlled trial. 70 participants will be recruited from the outpatient clinic of the department of Physical Medicine and Rehabilitation of Shin Kong Wu Ho-Su Memorial Hospital and randomly divided into COMB group and PT group. Each subject in the COMB group will receive 2 times of ultrasound-guided hydrodilatation injection (10mg triamcilonone, 2cc 1% xylocain, and 17cc normal saline) through both anterior and posterior shoulder joint in a two-weekly interval. In addition, joint mobilization and general physiotherapy (stretch exercise and physical modalities) will also be given, 2 times a week, for 8 weeks. The PT group will receive general physical therapy, 2 times a week, for 8 weeks. Outcome measures include the Shoulder Pain and Disability Index (SPADI), the Shoulder Disability Questionnaire (SDQ), and active and passive range of motion (ROM) of the affected shoulder, the 36-item Short Form Health Survey (SF-36), and patients' self evaluation. Evaluation will be performed at baseline and at 2, 4, 6 months after the beginning of the treatment. Statistics will be performed after completing the patients' treatment and evaluations. We expect that the COMB group will recover sooner and better than the PT group.

ELIGIBILITY:
Inclusion Criteria:

1. . age between 20 to 80 years old;
2. . chronic shoulder pain for ≥ 3 months;
3. . > 30% loss of passive range of motion (ROM) of the affected shoulder in either external rotation or abduction, comparing with the sound side;
4. . visual analog scale for pain on maximal passive external rotation or abduction > 4.

Exclusion Criteria:

1. . Severe systemic disorders including cancer, stroke, or cardiopulmonary diseases;
2. . Uncontrolled DM;
3. . Rotator cuff tear or calcification of the affected shoulder;
4. . Fracture, dislocation, or arthritis of the shoulder due to rheumatic disorders;
5. . a history of drug allergy to local anesthetics or corticosteroids;
6. . receiving corticosteroid or hyaluronic acid joint or bursa injection of the affected shoulder during the preceding three months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index（SPADI） | change between baseline and at 2 months, 4 months, 6 months after the beginning of the treatment.

SECONDARY OUTCOMES:
Visual analog scale（VAS） | change between baseline and at 2 months, 4 months, 6 months after the beginning of the treatment.
  The VAS for pain is obtained using a 100-mm-long horizontal line, with 0 mm on the left, indicating no pain, and 100 mm on the right, indicating very severe pain. The pain at rest is defined as rest pain, and pain on maximal abduction of the affected shoulder is defined as activity pain. The reliability of VAS for pain is 0.94, but in the absence of a criterion standard for pain, criterion validity cannot be evaluated.
Range of motion（ROM） | change between baseline and at 2 months, 4 months, 6 months after the beginning of the treatment.
  All the 4 planes of ROM will be measured. It includes abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 0° of abduction.
Shoulder Disability Questionnaire（SDQ） | change between baseline and at 2 months, 4 months, 6 months after the beginning of the treatment.
  The SDQ is a pain-related questionnaire that contains 16 items describing common situations that may induce symptoms in patients with shoulder disorders. The response options are "yes," "no," and "not applicable." The final score is calculated by dividing the number of positively scored items by the total number of applicable items and then multiplying this number by 100, which results in a final score ranging between 0 (no disability) and 100 (the worst possible condition).
The 36-item Short Form Health Survey（SF-36） | change between baseline and at 2 months, 4 months, 6 months after the beginning of the treatment.
  The SF-36 is a generic measure of quality of life and is composed of 8 subscales related to the following components: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each subscale generates a score from 0 to 100, and higher scores indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan